CLINICAL TRIAL: NCT05470634
Title: Trail-running après Arthroplastie du Genou ou de la Hanche/Trail-running After Knee or Hip Arthroplasty
Brief Title: Trail-running After Knee or Hip Arthroplasty
Acronym: TAKOHA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/CHU/14
Record Dates: First submitted 2022-07-18; First posted 2022-07-22 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-07

CONDITIONS: Arthropathy of Knee; Arthropathy of Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of indications for hip and knee arthroplasty is constantly increasing due to an increase in arthrogenic risk factors and life expectancy.

In younger patients, with a higher functional demand, resumption of physical activity and sport is a major objective after resumption of walking and pain management.

The repercussions of returning to sports after arthroplasty have been widely studied in the literature.

Few studies have looked specifically at high-impact activities, the possibility of resuming sport and its consequences. The recommendations are essentially based on expert opinion.

DETAILED DESCRIPTION:
The incidence of indications for hip and knee arthroplasty is constantly increasing due to an increase in arthrogenic risk factors and life expectancy. Projections predict an increase in the number of prosthetic surgeries between 2020 and 2030 of 150% for total hip replacements (THR) and 230% for total knee replacements (TKR).

In younger patients, with a higher functional demand, resumption of physical activity and sport is a major objective after resumption of walking and pain management. They are also more likely to resume physical activities with high peak joint stresses, known as "high-impact sports", most often against the advice of their surgeon.

The repercussions of returning to sports after arthroplasty have been widely studied in the literature. These are essentially descriptive cross-sectional studies which show greater participation in low or medium impact sports activities in patients with prostheses.

Few studies have looked specifically at high-impact activities, the possibility of resuming sport and its consequences. The recommendations are essentially based on expert opinion.

Concerning trail running, a discipline in full expansion, particularly in the longest formats; a single study in 2019, involving 18 runners with a prosthesis, did not reveal any specific constraints compared to healthy runners during a 170 km ultratrail.

ELIGIBILITY:
Inclusion Criteria:

* Trail runner (declarative)
* Having been operated for a hip or knee arthroplasty
* No limit to the length of time or volume of trail riding

Exclusion Criteria:

* Refusal to participate
* Trailer not understanding French

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The recruitment process will involve a pre-recruitment informing runners that we are looking for trail runners of all levels who have undergone hip and knee replacement surgery. This information will be disseminated via social networks, trail clubs, and via the organisers of major trail races (Diagonale des Fous, UTMB). We will then send the questionnaires to all the runners who have replied to us and mentioned their willingness to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
To evaluate the impact of trail running on patients who have undergone prosthetic surgery (total or partial hip or knee arthroplasty) on the quality of life | Day 1
  This impact will be assessed using :
  -the EuroQol Group 5D-5L (EQ5D-5L) score (with 0 being yhe worst score and 100 the best score)
To evaluate the impact of trail running on patients who have undergone prosthetic surgery (total or partial hip or knee arthroplasty) on physical activity | Day 1
  This impact will be assessed using :
  - UCLA (University of California, Los Angeles) score 10 (ranging from wholly inactive and dependent (level 1) to regular participation in impact sports (level 10))
To evaluate the impact of trail running on patients who have undergone prosthetic surgery (total or partial hip or knee arthroplasty) on hip problems | Day 1
  This impact will be assessed using :
  - the HOOS12 scale (Hip and Osteoarthritis Outcome Score) with 12 questions scored from 1 to 4 each, with 0 representing no hip problems and 4 representing extreme hip problems
To evaluate the impact of trail running on patients who have undergone prosthetic surgery (total or partial hip or knee arthroplasty) on knee problems | Day 1
  This impact will be assessed using :
  - KOOS12 scale (Knee and Osteoarthritis Outcome Score) with 12 questions scored from 1 to 4 each, with 0 representing no knee problems and 4 representing extreme knee problems

SECONDARY OUTCOMES:
Functional scores of the hip and knee prostheses | Day 1
  Compare the functional scores of the hip and knee prostheses of these patients using the HOOS12 scale (Hip and Osteoarthritis Outcome Score) with 12 questions scored from 1 to 4 each, with 0 representing no hip problems and 4 representing extreme hip problems and the KOOS12 scale (Knee and Osteoarthritis Outcome Score) with 12 questions scored from 1 to 4 each, with 0 representing no knee problems and 4 representing extreme knee problems
Pain and satisfactory level | Day 1
  Evaluate the pain and satisfaction of these patients after returning to running after a prosthetic surgery using the study questionnaire
Rehabilitation and physical preparation | Day 1
  To analyse the rehabilitation and physical preparation of these patients that allowed them to return to sport after hip and knee prothesis implantation using the study questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Cédric MAILLOT, MD, Principal Investigator — CHU La Réunion
Locations (1):
- CHU de la Réunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No